CLINICAL TRIAL: NCT04594252
Title: A Phase 1, Open-label Study to Assess Copper Balance in Healthy Participants Following Administration of ALXN1840
Brief Title: Copper Balance in Healthy Participants Administered ALXN1840
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1840-HV-108
Record Dates: First submitted 2020-09-28; First posted 2020-10-20 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Copper Balance; Molybdenum Balance; Healthy; ALXN1840

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN1840 (Experimental): Participants will be administered repeat doses of ALXN1840 30 milligrams (mg) for 15 days.
  Interventions: Drug: ALXN1840

INTERVENTIONS:
Drug: ALXN1840 — Administered orally as tablets.
  Other Names: formerly WTX101

SUMMARY:
The study will assess the change from baseline in mean daily copper balance in healthy participants with repeat-dose administrations of ALXN1840 over 2 weeks.

DETAILED DESCRIPTION:
This study will also characterize the steady state absorption, distribution, metabolism, and excretion (mass balance) of total molybdenum, which is a surrogate measure of ALXN1840 disposition.

Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have regular bowel movements (at least once per day).
2. Adequate venous access in the left or right arm to allow collection of study-required blood samples.
3. Willing and able to adhere to all dietary requirements of the study.
4. Body weight between 50 to 70 kilograms (kg) (inclusive) for female participants, and 65 to 85 kg (inclusive) for male participants, and body mass index within the range 18 to 25 kg/meters squared (inclusive).
5. Willing and able to follow protocol-specified contraception requirements.
6. Capable of giving signed informed consent.

Exclusion Criteria:

1. Significant medical history (current or past).
2. History or presence of gastrointestinal conditions including chronic constipation and irritable bowel syndrome.
3. Supine blood pressure ≤ 90/60 millimeters of mercury (mmHg) or > 140/90 mmHg.
4. Lymphoma, leukemia, or any malignancy within 3 years.
5. Breast cancer within the past 10 years.
6. Alanine aminotransferase, aspartate aminotransferase, or total bilirubin > upper limit of normal at Screening.
7. Serum copper or serum ceruloplasmin below lower limit of normal on laboratory reference range at Screening.
8. History of anemia or hemoglobin < 130 gram (g)/Liter (L) for men and hemoglobin < 115 g/L for women at Screening.
9. History of benign ethnic neutropenia or absolute neutrophil count < 1500/microliter (uL), lymphocyte count below 1000/uL.
10. QTcF> 450 millisecond (ms) for men and QTcF> 480 ms for women.
11. Current or chronic history of liver disease or known hepatic or biliary abnormalities (except for asymptomatic gallstones).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.; Peter Ksenuk, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (1):
- Clinical Study Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 17 participants were enrolled in 2 groups. Group 1 consisted of 6 participants. Group 2, consisting of 11 participants, was initiated after the Safety Review Committee (SRC) reviewed safety information from Group 1. No safety concerns were identified; therefore, no dose adjustments were implemented with Group 2.
Groups:
- Group 1: ALXN1840; Group 2: ALXN1840: Participants received repeat dose of ALXN1840 tablet administered orally on Day 1 through Day 15.
Period: Overall Study
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840
Started | 6 | 11
Received at Least 1 Dose of Study Drug | 6 | 11
Completed | 6 | 9
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (6.29) | 29.5 (5.61) | 28.6 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mean Daily Copper Balance [Mean (Standard Deviation); unit: milligrams (mg)/day] | 0.8538 (0.48629) | 0.3317 (0.44568) | 0.5160 (0.51399)
Mean Daily Molybdenum Balance [Mean (Standard Deviation); unit: mg/day] | 0.1286 (0.04469) | 0.0133 (0.05035) | 0.0540 (0.07372)
Total Molybdenum Excretion in Feces [Mean (Standard Deviation); unit: mg] | 0.0586 (0.02347) | 0.0724 (0.03023) | 0.0675 (0.02809)
Total Molybdenum Excretion in Urine [Mean (Standard Deviation); unit: mg] | 0.1039 (0.02656) | 0.1198 (0.03546) | 0.1142 (0.03268)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daily Copper Balance Over 2 Weeks of Repeated Daily ALXN1840 Dosing (Over Days 4 to 15)
Description: Copper balance was defined as the difference in copper input and copper output. A negative copper balance indicated greater copper output than copper intake. Copper input was defined as the sum of all copper input as measured in all food and fluids over the specified period. Copper output was defined as the sum of all copper output as measured in urine and feces over the specified collection period. Baseline was defined as the average of the nonmissing values on or before first study drug administration from Day -4 to Day -1.
Time Frame: Baseline, Days 4 to 15
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg/day
Groups:
- Total (Groups 1 and 2): ALXN1840: Participants received repeat dose of ALXN1840 tablet administered orally on Day 1 through Day 15.
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg/day | -0.0749 (0.37419) | 0.6901 (0.48176) | 0.4201 (0.57518)

2. Secondary Outcome: Mean Daily Copper Balance Over Two Weeks of Repeated ALXN1840 Dosing
Description: Copper balance was defined by the difference in copper input and copper output. A negative copper balance indicated greater copper output than copper intake. Copper input was defined as the sum of all copper input as measured in all food and fluids over the specified period. Copper output was defined as the sum of all copper output as measured in urine and feces over the specified collection period.
Time Frame: Day 4 through Day 15
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg/day | 0.7789 (0.20297) | 1.0218 (0.21279) | 0.9361 (0.23558)

3. Secondary Outcome: Change From Baseline in Mean Daily Molybdenum Balance at Steady State (Over Days 12 to 15)
Description: Molybdenum mass balance was defined as the difference in molybdenum input and molybdenum output. A negative molybdenum balance indicated greater molybdenum output than molybdenum intake. Molybdenum input was defined as the sum of all molybdenum input as measured in all food and fluids over the specified period. Molybdenum output was defined as the sum of all molybdenum output as measured in urine and feces over the specified collection period. Baseline was defined as the average of the nonmissing values on or before first study drug administration from Day -4 to Day -1.
Time Frame: Baseline, Days 12 to 15
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg/day | 1.7750 (0.98161) | 0.6189 (1.24337) | 1.0269 (1.26161)

4. Secondary Outcome: Change From Baseline in Total Molybdenum Excretion in Urine and Feces Averaged Over 2 Weeks of Dosing (Days 4 to 15)
Description: Molybdenum mass balance was defined as the difference in molybdenum input and molybdenum output. A negative molybdenum balance indicated greater molybdenum output than molybdenum intake. Molybdenum input was defined as the sum of all molybdenum input as measured in all food and fluids over the specified period. Molybdenum output was defined as the sum of all molybdenum output as measured in urine and feces over the specified collection period. Baseline was defined as the average of the nonmissing values on or before first study drug administration from Day -4 to Day -1. Molybdenum excretion for the Day 4 through Day 15 period included data averaged from Day 4 through Day 15.
Time Frame: Baseline, Days 4 to 15
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg
  Urine | 2.6210 (0.68681) | 2.5957 (0.39688) | 2.6046 (0.49600)
  Feces | 2.0247 (0.64199) | 1.9586 (0.32854) | 1.9819 (0.44421)

5. Secondary Outcome: Mean Daily Molybdenum Balance Throughout the ALXN1840 Treatment Period (Day 1 Through Day 15)
Description: Molybdenum mass balance was defined as the difference in molybdenum input and molybdenum output. A negative molybdenum balance indicated greater molybdenum output than molybdenum intake. Molybdenum input was defined as the sum of all molybdenum input as measured in all food and fluids over the specified period. Molybdenum output was defined as the sum of all molybdenum output as measured in urine and feces over the specified collection period.
Time Frame: Day 1 through Day 15
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg/day | 2.5560 (0.73042) | 2.2861 (0.35654) | 2.3813 (0.51367)

6. Secondary Outcome: Copper Quantified in Food, Drink, Feces, and Urine Averaged Over 2 Weeks of Dosing
Description: Copper balance for the Day 4 through Day 15 period included data averaged from Day 4 through Day 15.
Time Frame: Days 4 to 15
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg
  Copper Quantified in Food | 1.5039 (0.10025) | 1.7178 (0.12247) | 1.6423 (0.15366)
  Copper Quantified in Drink | 0.0270 (0.00120) | 0.0108 (0.00194) | 0.0165 (0.00816)
  Copper Quantified in Feces | 0.7373 (0.23986) | 0.6895 (0.17102) | 0.7064 (0.19187)
  Copper Quantified in Urine | 0.0147 (0.01102) | 0.0173 (0.00780) | 0.0164 (0.00881)

7. Secondary Outcome: Copper Quantified in Food, Drink, Feces, and Urine From Day 1 Through Day 30
Description: Copper balance for the Day 1 through Day 30 period included data averaged from Day 1 through Day 30.
Time Frame: Day 1 through Day 30
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg
  Copper Quantified in Food | 1.6117 (0.12736) | 1.6673 (0.12779) | 1.6476 (0.12659)
  Copper Quantified in Drink | 0.0252 (0.00124) | 0.0124 (0.00212) | 0.0169 (0.00658)
  Copper Quantified in Feces | 0.7017 (0.19009) | 0.6962 (0.13385) | 0.6982 (0.14999)
  Copper Quantified in Urine | 0.0192 (0.01107) | 0.0209 (0.00655) | 0.0203 (0.00811)

8. Secondary Outcome: Plasma Total Copper Concentration and Labile Bound Copper (LBC) Concentration
Time Frame: Day 15 (predose and 24 hours postdose)
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840. Here, 'number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: micromoles (μmol)/liter (L)
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
micromoles (μmol)/liter (L)
  Total Copper Concentration at Day 15 (predose) | 12.58931 (1.636640) | 13.87256 (1.627496) | 13.41964 (1.700617)
  Total Copper Concentration at Day 15 (24 hours postdose): number analyzed (Participants) | 6 | 10 | 16
  Total Copper Concentration at Day 15 (24 hours postdose) | 12.56570 (1.342502) | 14.49816 (1.548441) | 13.77349 (1.724230)
  LBC Concentration at Day 15 (predose) | 0.93213 (0.262655) | 0.82360 (0.160887) | 0.86190 (0.201482)
  LBC Concentration at Day 15 (24 hours postdose): number analyzed (Participants) | 6 | 10 | 16
  LBC Concentration at Day 15 (24 hours postdose) | 1.04386 (0.233526) | 0.90612 (0.264791) | 0.95777 (0.254932)

9. Secondary Outcome: Molybdenum Quantified in ALXN1840 Doses Given and in Food, Drink, Feces, And Urine
Description: Molybdenum balance for the Day 1 through Day 30 period included data averaged from Day 1 through Day 30.
Time Frame: Day 1 through Day 30
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
mg
  Molybdenum Quantified in Food | 0.2618 (0.02275) | 0.1414 (0.01123) | 0.1839 (0.06129)
  Molybdenum Quantified in Drink | 0.0014 (0.00015) | 0.0017 (0.00048) | 0.0016 (0.00041)
  Molybdenum Quantified in Feces | 1.0575 (0.29359) | 0.9949 (0.16082) | 1.0170 (0.20988)
  Molybdenum Quantified in Urine | 1.4016 (0.35415) | 1.3848 (0.21874) | 1.3907 (0.26300)
  Molybdenum Quantified in ALXN1840 Doses Given | 3.5933 (0.02277) | 3.3625 (0.28101) | 3.4439 (0.24988)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Molybdenum and Plasma Ultrafiltrate (PUF) Molybdenum
Time Frame: Predose (within 1 hour prior to dosing) through 24 hours postdose on Day 1 and Day 15
Population: Pharmacokinetic (PK) analysis set included all participants who had sufficient samples to enable the calculation of PK parameters and provide PK profiles. Here, 'number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
nanograms (ng)/mL
  Cmax of Total Molybdenum at Day 1 | 303.000 (65.3667) | 291.727 (100.7324) | 295.706 (87.7950)
  Cmax of Total Molybdenum at Day 15: number analyzed (Participants) | 6 | 9 | 15
  Cmax of Total Molybdenum at Day 15 | 358.500 (53.6945) | 382.333 (78.2624) | 372.800 (68.3794)
  Cmax of PUF Molybdenum at Day 1 | 30.445 (12.0613) | 27.266 (12.9396) | 28.388 (12.3515)
  Cmax of PUF Molybdenum at Day 15: number analyzed (Participants) | 6 | 9 | 15
  Cmax of PUF Molybdenum at Day 15 | 93.717 (42.9368) | 74.678 (36.1617) | 82.293 (38.7152)

11. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval (AUCtau) of Total Molybdenum and PUF Molybdenum
Time Frame: Predose (within 1 hour prior to dosing) through 24 hours postdose on Day 1 and Day 15
Population: PK analysis set included all participants who had sufficient samples to enable the calculation of PK parameters and provide PK profiles. Here, 'number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
hours*ng/mL
  AUCtau of Total Molybdenum at Day 1 | 4860.289 (1078.263) | 4439.012 (1374.869) | 4587.698 (1260.082)
  AUCtau of Total Molybdenum at Day 15: number analyzed (Participants) | 6 | 9 | 15
  AUCtau of Total Molybdenum at Day 15 | 6770.905 (582.770) | 7496.724 (1499.370) | 7206.397 (1241.529)
  AUCtau of PUF Molybdenum at Day 1 | 356.156 (133.8174) | 318.123 (131.9084) | 331.546 (129.6990)
  AUCtau of PUF Molybdenum at Day 15: number analyzed (Participants) | 6 | 9 | 15
  AUCtau of PUF Molybdenum at Day 15 | 1035.231 (252.0931) | 913.807 (379.1750) | 962.376 (329.6126)

12. Secondary Outcome: Observed Concentration at the End of the Dosing Interval (Ctau) of Total Molybdenum and PUF Molybdenum
Time Frame: Predose (within 1 hour prior to dosing) through 24 hours postdose on Day 1 and Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
Number analyzed (Participants) | 6 | 11 | 17
ng/mL
  Ctau of Total Molybdenum at Day 1 | 143.800 (35.5348) | 140.436 (53.2088) | 141.624 (46.5492)
  Ctau of Total Molybdenum at Day 15: number analyzed (Participants) | 6 | 8 | 14
  Ctau of Total Molybdenum at Day 15 | 218.833 (23.0340) | 242.625 (54.5892) | 232.429 (44.2488)
  Ctau of PUF Molybdenum at Day 1 | 4.655 (1.1623) | 4.785 (1.6602) | 4.739 (1.4660)
  Ctau of PUF Molybdenum at Day 15: number analyzed (Participants) | 6 | 8 | 14
  Ctau of PUF Molybdenum at Day 15 | 11.060 (1.3785) | 11.141 (2.8492) | 11.106 (2.2591)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 43
Description: Safety set included all participants who received at least 1 dose of ALXN1840.
Arm/Group | Group 1: ALXN1840 | Group 2: ALXN1840 | Total (Groups 1 and 2): ALXN1840
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 5/6 | 9/11 | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: ALXN1840 (N=6) | Group 2: ALXN1840 (N=11) | Total (Groups 1 and 2): ALXN1840 (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 3 (4)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2/3 (2) | 0/6 (0) | 2/9 (2) — This is a gender-specific AE. Only female participants were at risk.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT04594252/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04594252/SAP_001.pdf